CLINICAL TRIAL: NCT03645460
Title: Gene Therapy Via Intravenous Injection of Lentiviral Vector (Ivlv-ADA) for the Treatment of Adenosine Deaminase-severe Combined Immunodeficiency (ADA-SCID)
Brief Title: Gene Therapy for ADA-SCID Using an Improved Lentiviral Vector (Ivlv-ADA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-18003
Record Dates: First submitted 2018-07-17; First posted 2018-08-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Adenosine DeAminase Severe Combined ImmunoDeficiency (ADA-SCID)
Keywords: Adenosine deaminase severe combined immunodeficiency lentiviral vector; in vivo gene therapy
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct intravenous injection of ivlv-ADA lentiviral vector (Experimental): Direct intravenous injection of ivlv-ADA lentiviral vector
  Interventions: Genetic: Direct intravenous injection of ivlv-ADA lentiviral vector

INTERVENTIONS:
Genetic: Direct intravenous injection of ivlv-ADA lentiviral vector — Injection of ivlv-ADA lentiviral vector at ~1x10^9 per kg body weight

SUMMARY:
This is a Phase I/II trial of in vivo lentiviral gene therapy for treating adenosine deaminase severe combined immunodeficiency (ADA-SCID) using a self-inactivating lentiviral vector (LV) ivlv-ADA to functionally correct the genetic defect. The primary objectives are to evaluate the safety and efficacy of the direct intravenous (iv) LV gene therapy protocol.

DETAILED DESCRIPTION:
This clinical trial will evaluate safety and efficiency of an improved LV system for delivering a therapeutic gene to patients with severe combined immunodeficiency (SCID) due to a defective adenosine deaminase (ADA) gene. This gene encodes for the adenosine deaminase enzyme, which is essential for the proper growth and function of infection-fighting white blood cells called T and B lymphocytes. Patients who lack this enzyme are vulnerable to frequent and severe infections.

ADA-SCID patients are normally rescued by a bone marrow transplant (BMT) from a matched healthy donor. However, matched donors are difficult to find and donor BMT is associated with high risk. This trial aims to treat ADA-SCID via direct intravenous (iv) injection of a safety and efficiency improved self-inactivating LV carrying a functional ADA gene (ivlv-ADA) to correct the genetic defect. By direct iv injection of ivlv-ADA, the defective immune cells and blood stem cells in the body can be modified to exhibit ADA activity and correct the immunodeficiency.

The primary objectives are to evaluate the safety of the improved ivlv-ADA, the iv LV gene transfer clinical protocol and the efficacy of immune recovery in patients to overcome frequent infections present at the time of treatment. We will assess the in vivo lentiviral gene transfer efficiency and the long-term effect of this gene transfer procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of classical ADA-SCID based on:

  * A proven defective adenosine deaminase (ADA) gene as defined by direct sequencing of patient DNA.
  * T-cell immune deficiency defined as one or more of the following: CD3+ autologous T cells < 300/ul, or less than 50% of normal value for in vitro mitogen stimulation, or absent proliferation in vitro to antigens.
* With severe infections, including but not limited to: pneumonitis; protracted diarrhea requiring total parenteral nutrition; infection with herpes viruses or adenovirus or fungus; disseminated BCG infection.
* No cytogenetic abnormalities (medullary karyotype) and no detection of main rearrangements associated with acute leukemia of children.
* No prior allogeneic stem cell transplantation.
* Life expectancy ≥ 2 months.
* Negative for HIV infection.
* Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

* None

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival up to a year | 1 years
  Patient will be monitored for overall health condition, including immune cell assessments, blood biochemistry and metabolitic activities, metabolic detoxification, gene-modified cell percentage and vector copy number (VCN) in the blood, and continued follow-up for 1 years.

SECONDARY OUTCOMES:
1. Success of immune reconstitution | 12 month
  Immunological and metabolic values including all leukocyte counts (ALC), T, B and NK cell counts (CD3, CD4, CD8, CD19, CD56), T cell TREC levels, T cell repertoire diversity, PHA proliferation rate, immunoglobulins and dATP levels will be measured.
2. Change of infection status | 12 month
  Immune recovery associated with reduction of infection episodes and frequencies, including viral, fungal and bacterial infections will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Ph.D, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (2):
- China (2):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Guilin Hospital of Chinese Traditional and Western Medicine, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No